CLINICAL TRIAL: NCT02601001
Title: A Phase 1, Single Center Double-blind, Randomized, Placebo-controlled Study to Evaluate the Pharmacokinetics and Safety of Omecamtiv Mecarbil in Healthy Japanese Subjects
Brief Title: Pharmacokinetics and Safety Study of Omecamtiv Mecarbil in Healthy Japanese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150134
Record Dates: First submitted 2015-06-17; First posted 2015-11-10 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteer
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received placebo tablets twice a day (BID) in dosing period 1 (days 1 to 8) and in dosing period 2 (days 20 to 27).
  Interventions: Drug: Placebo
- Omecamtiv mecarbil 25 mg / 37.5 mg (Experimental): Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 25 mg or 37.5 mg BID in dosing period 2 (days 20 to 27) based on their day 8 predose omecamtiv mecarbil plasma concentration (Cpredose): If day 8 Cpredose was < 200 ng/mL, participants received 37.5 mg BID; if day 8 Cpredose was ≥ 200 ng/mL or a day 8 PK value was not available participants continued to receive 25 mg BID.
  Interventions: Drug: Omecamtiv mecarbil
- Omecamtiv mecarbil 25 mg / 50 mg (Experimental): Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 25 mg or 50 mg BID in dosing period 2 (days 20 to 27) based on their day 8 predose omecamtiv mecarbil plasma concentration (Cpredose): If day 8 Cpredose was < 200 ng/mL, participants received 50 mg BID; if day 8 Cpredose was ≥ 200 ng/mL or a day 8 PK value was not available participants continued to receive 25 mg BID.
  Interventions: Drug: Omecamtiv mecarbil

INTERVENTIONS:
Drug: Omecamtiv mecarbil — Omecamtiv mecarbil tablets for oral administration
  Other Names: AMG 423
  Arms: Omecamtiv mecarbil 25 mg / 37.5 mg; Omecamtiv mecarbil 25 mg / 50 mg
Drug: Placebo — Matching placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of omecamtiv mecarbil in healthy volunteers in Japan.

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* No history or evidence of clinically relevant medical disorders as determined by the Investigator, and in good health as determined by a pre-study physical examination and medical history with no clinically significant abnormalities, normal vital signs and no history or presence of a clinically significant abnormal electrocardiogram finding
* Subjects' pre-study clinical laboratory findings (including creatine phosphokinase) should be within normal range or if outside of the normal range, are deemed not clinically significant by the Investigator.

Exclusion Criteria:

* A clinically significant disorder/disease, including gastro intestinal abnormalities that might interfere with absorption
* An unstable medical condition, defined as having been hospitalized within 28 days before day 1, major surgery within 6 months before day 1, or otherwise unstable in the judgment of the Investigator
* History or evidence of any other clinically significant disorder, condition, or disease that, in the opinion of the Investigator or Medical Monitor would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* History of malignancy of any type other than surgically excised non-melanomatous skin cancers or in situ cervical cancer within 5 years before the day of dosing
* Use of any prescription or over-the-counter medications within 14 days or 5 half-lives (whichever time period is greater), prior to receiving the first dose of omecamtiv mecarbil (acetaminophen up to 2 grams per day for analgesia and hormone replacement therapy (e.g., estrogen) will be allowed
* Use of any known inhibitors of CYP3A4/p-glycoprotein (P-gp) or CYP2D6 within 14 days or 5 half-lives, whichever is longer; or use of grapefruit juice or grapefruit containing products within 7 days prior to receiving the first dose of omecamtiv mecarbil
* Use of any known CYP3A4 inducers within 30 days or 5 half-lives, whichever is longer, before receiving omecamtiv mecarbil

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-13 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2016-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Kagoshima, Kagoshima-ken, Japan

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in Japan. Participants were enrolled from 13 November 2015 to 24 November 2015.
Pre-assignment Details: Participants were randomly assigned to one of three treatment groups in a 1:2:2 ratio.
  The study consisted of a screening period, two 8-day treatment periods with an 11-day drug holiday in between, and an end of study (EOS) visit on day 35.
Groups:
- Period 1 Group A: Omecamtiv Mecarbil 25 mg: Participants received omecamtiv mecarbil (OM) 25 mg BID in dosing period 1 (days 1 to 8).
- Period 1 Group B: Omecamtiv Mecarbil 25 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8).
- Period 2 Group A: Omecamtiv Mecarbil 25 mg: Participants who received omecamtiv mecarbil 25 mg BID in dosing period 1 then received omecamtiv mecarbil 25 mg BID in dosing period 2 (days 20 to 27) based on their day 8 predose omecamtiv mecarbil plasma concentration (Cpredose).
- Period 2 Group A: Omecamtiv Mecarbil 37.5 mg: Participants who received omecamtiv mecarbil 25 mg BID in dosing period 1 then received omecamtiv mecarbil 37.5 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Period 2 Group B: Omecamtiv Mecarbil 25 mg: Participants who received omecamtiv mecarbil 25 mg BID in dosing period 1 then received omecamtiv mecarbil 25 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Period 2 Group B: Omecamtiv Mecarbil 50 mg: Participants who received omecamtiv mecarbil 25 mg BID in dosing period 1 then received omecamtiv mecarbil 50 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
Period: Dosing Period 1
Arm/Group | Placebo | Period 1 Group A: Omecamtiv Mecarbil 25 mg | Period 1 Group B: Omecamtiv Mecarbil 25 mg | Period 2 Group A: Omecamtiv Mecarbil 25 mg | Period 2 Group A: Omecamtiv Mecarbil 37.5 mg | Period 2 Group B: Omecamtiv Mecarbil 25 mg | Period 2 Group B: Omecamtiv Mecarbil 50 mg
Started | 10 | 20 | 20 | 0 | 0 | 0 | 0
Completed (Completed dosing in period 1) | 10 | 20 | 20 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dosing Period 2
Arm/Group | Placebo | Period 1 Group A: Omecamtiv Mecarbil 25 mg | Period 1 Group B: Omecamtiv Mecarbil 25 mg | Period 2 Group A: Omecamtiv Mecarbil 25 mg | Period 2 Group A: Omecamtiv Mecarbil 37.5 mg | Period 2 Group B: Omecamtiv Mecarbil 25 mg | Period 2 Group B: Omecamtiv Mecarbil 50 mg
Started | 10 | 0 | 0 | 7 | 13 | 7 | 13
Completed (Completed dosing in period 2) | 10 | 0 | 0 | 7 | 13 | 7 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 25 mg or 37.5 mg BID in dosing period 2 (days 20 to 27) based on their day 8 predose omecamtiv mecarbil plasma concentration (Cpredose): If day 8 Cpredose was < 200 ng/mL, participants received 37.5 mg BID; if day 8 Cpredose was ≥ 200 ng/mL participants continued to receive 25 mg BID.
- Group B: Omecamtiv Mecarbil 25 mg / 50 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 25 mg or 50 mg BID in dosing period 2 (days 20 to 27) based on their day 8 predose omecamtiv mecarbil plasma concentration (Cpredose): If day 8 Cpredose was < 200 ng/mL, participants received 50 mg BID; if day 8 Cpredose was ≥ 200 ng/mL participants continued to receive 25 mg BID.
- Total: Total of all reporting groups
Arm/Group | Placebo | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg | Total
Number analyzed (Participants) | 10 | 20 | 20 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.2) | 35.5 (7.6) | 27.3 (4.6) | 31.0 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 6 | 15
  Male | 7 | 14 | 14 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 20 | 20 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 20 | 20 | 50
  Black or African American | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Dosing Period 1: Maximum Observed Plasma Concentration (Cmax) of Omecamtiv Mecarbil After First and Last Dose in Period 1
Time Frame: Day 1 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose. Day 8 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours after the morning dose.
Population: The pharmacokinetic (PK) analysis set included all randomized participants who received at least 1 dose of omecamtiv mecarbil and had at least 1 evaluable omecamtiv mecarbil PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group A: Omecamtiv Mecarbil 25 mg; Group B: Omecamtiv Mecarbil 25 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8).
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg | Group B: Omecamtiv Mecarbil 25 mg
Number analyzed (Participants) | 20 | 20
ng/mL
  After first dose on day 1 | 77.4 (21.6) | 79.5 (18.9)
  After last dose on day 8 | 256 (71.2) | 259 (59.2)

2. Primary Outcome: Dosing Period 1: Time to Maximum Observed Plasma Concentration (Tmax) of Omecamtiv Mecarbil After First and Last Dose in Period 1
Time Frame: as for outcome 1
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg | Group B: Omecamtiv Mecarbil 25 mg
Number analyzed (Participants) | 20 | 20
hours
  After first dose on day 1 | 4.0 [0.5 to 8.0] | 3.0 [0.5 to 8.0]
  After last dose on day 8 | 2.0 [0.5 to 4.0] | 2.0 [0.5 to 8.0]

3. Primary Outcome: Dosing Period 1: Area Under the Concentration-time Curve for a Dosing Interval of 12 Hours (AUC0-12) for Omecamtiv Mecarbil After First and Last Dose in Period 1
Time Frame: Day 1 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose. Day 8 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose.
Population: The PK analysis set with available AUC data at each time point
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg | Group B: Omecamtiv Mecarbil 25 mg
Number analyzed (Participants) | 20 | 20
ng*hr/mL
  After first dose on day 1: number analyzed (Participants) | 10 | 14
  After first dose on day 1 | 687 (210) | 677 (163)
  After last dose on day 8 | 2570 (739) | 2670 (699)

4. Primary Outcome: Dosing Period 1: Predose Omecamtiv Mecarbil Plasma Concentration
Time Frame: Day 8 predose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg | Group B: Omecamtiv Mecarbil 25 mg
Number analyzed (Participants) | 20 | 20
ng/mL | 190 (58.5) | 192 (55.1)

5. Primary Outcome: Dosing Period 1: Accumulation Ratio
Description: Accumulation ratio calculated as the ratio of day 8 AUC(0-12) / day 1 AUC(0-12)
Time Frame: as for outcome 3
Population: The PK analysis set with available AUC data at both time points
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg | Group B: Omecamtiv Mecarbil 25 mg
Number analyzed (Participants) | 10 | 14
ratio | 3.66 (0.89) | 3.79 (0.77)

6. Primary Outcome: Dosing Period 2: Maximum Observed Plasma Concentration (Cmax) of Omecamtiv Mecarbil After First and Last Dose in Period 2
Time Frame: Day 20 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose. Day 27 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours after the morning dose.
Population: Pharmacokinetic analysis set with available data at each time point
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Group A: Omecamtiv Mecarbil 25 mg / 25 mg; Group B: Omecamtiv Mecarbil 25 mg / 25 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 25 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 37.5 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Group B: Omecamtiv Mecarbil 25 mg / 50 mg: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8) and 50 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 7 | 13 | 7 | 13
ng/mL
  After first dose on day 20 | 96.5 (27.2) | 107 (30.4) | 84.9 (30.0) | 154 (22.0)
  After last dose on day 27: number analyzed (Participants) | 7 | 13 | 7 | 12
  After last dose on day 27 | 335 (32.0) | 341 (48.8) | 311 (54.2) | 537 (91.7)

7. Primary Outcome: Dosing Period 2: Time to Maximum Observed Plasma Concentration (Tmax) of Omecamtiv Mecarbil After First and Last Dose in Period 2
Time Frame: as for outcome 6
Population: Pharmacokinetic analysis set with available data at each time point
Measure: Median (Full Range); unit: hours
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 7 | 13 | 7 | 13
hours
  After first dose on day 20 | 4.0 [2.0 to 11] | 2.0 [0.5 to 6.0] | 4.0 [1.0 to 11] | 3.0 [0.5 to 6.0]
  After last dose on day 27: number analyzed (Participants) | 7 | 13 | 7 | 12
  After last dose on day 27 | 2.0 [0.5 to 4.0] | 3.0 [0.5 to 4.0] | 4.0 [0.5 to 4.0] | 3.0 [0.5 to 4.0]

8. Primary Outcome: Dosing Period 2: AUC(0-12) for Omecamtiv Mecarbil After First and Last Dose in Period 2
Time Frame: Day 20 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose. Day 27 at 0 hours and 0.5, 1, 2, 3, 4, 6, 8, and 12 hours after the morning dose.
Population: Pharmacokinetic analysis set with available AUC data at each time point
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 7 | 13 | 7 | 13
ng*hr/mL
  After first dose on day 20: number analyzed (Participants) | 4 | 10 | 4 | 10
  After first dose on day 20 | 902 (220) | 950 (228) | 841 (403) | 1330 (217)
  After last dose on day 27: number analyzed (Participants) | 7 | 13 | 7 | 12
  After last dose on day 27 | 3520 (505) | 3500 (519) | 3290 (662) | 5490 (1000)

9. Primary Outcome: Dosing Period 2: Predose Omecamtiv Mecarbil Plasma Concentration
Time Frame: Day 27 predose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 7 | 13 | 7 | 12
ng/mL | 271 (44.8) | 256 (42.1) | 245 (43.3) | 401 (77.8)

10. Primary Outcome: Dosing Period 2: Accumulation Ratio
Description: Accumulation ratio calculated as the ratio of day 27 AUC(0-12) / day 20 AUC(0-12).
Time Frame: as for outcome 8
Population: Pharmacokinetic analysis set with available AUC data at both time points
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 4 | 10 | 4 | 9
ratio | 4.12 (1.28) | 3.81 (0.83) | 4.53 (1.19) | 4.11 (1.15)

11. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An adverse event is defined as any untoward medical occurrence in a clinical trial participant, including worsening of a preexisting medical condition. The event does not necessarily have a causal relationship with study treatment.
  A serious adverse event is defined as an adverse event that met at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * required in patient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. Adverse events were graded for severity according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 35 days
Population: All randomized participants who received at least one dose of study treatment (omecamtiv mecarbil or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 10 | 7 | 13 | 7 | 13
Participants
  Any treatment-emergent adverse event | 6 | 4 | 7 | 4 | 3
  Serious adverse events | 0 | 0 | 0 | 0 | 0
  TEAE leading to discontinuation of study drug | 0 | 0 | 0 | 0 | 1
  Severe adverse events | 0 | 0 | 0 | 1 | 1
  Life-threatening adverse events | 0 | 0 | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Grade 3 or Higher Laboratory Toxicities
Description: Abnormal laboratory findings were graded for severity according to the NCI CTCAE version 4.0 according to the following guideline:
  * Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  * Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL).
  * Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL.
  * Grade 4: Life-threatening consequences; urgent intervention indicated.
  * Grade 5: Death related to AE.
Time Frame: 35 days
Population: All randomized participants who received at least one dose of study treatment (omecamtiv mecarbil or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 10 | 7 | 13 | 7 | 13
Participants | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Maximum Increase From Baseline in Fridericia-Corrected QT Interval (QTcF) In Dosing Period 1
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle as measured by electrocardiogram (ECG).
  Maximum increase from Period 1 baseline was categorized as:
  ≤ 30 milliseconds (ms) > 30 to 60 ms > 60 ms
Time Frame: Day 1 predose and day 8
Population: All randomized participants who received at least one dose of study treatment (omecamtiv mecarbil or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 10 | 7 | 13 | 7 | 13
Participants
  ≤ 30 ms | 10 | 7 | 13 | 7 | 13
  > 30 to 60 ms | 0 | 0 | 0 | 0 | 0
  > 60 ms | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Maximum Increase From Baseline in Fridericia-Corrected QT Interval (QTcF) In Dosing Period 2
Description: QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle as measured by ECG.
  Maximum increase from Period 2 baseline was categorized as:
  ≤ 30 ms > 30 to 60 ms > 60 ms
Time Frame: Day 20 predose and Day 27
Population: Randomized participants who received at least one dose of study treatment (omecamtiv mecarbil or placebo), with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Group A: Omecamtiv Mecarbil 25 mg / 25 mg | Group A: Omecamtiv Mecarbil 25 mg / 37.5 mg | Group B: Omecamtiv Mecarbil 25 mg / 25 mg | Group B: Omecamtiv Mecarbil 25 mg / 50 mg
Number analyzed (Participants) | 10 | 7 | 13 | 7 | 12
Participants
  ≤ 30 ms | 10 | 7 | 13 | 7 | 12
  > 30 to 60 ms | 0 | 0 | 0 | 0 | 0
  > 60 ms | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Period 1: Day 1 to day 19 Period 2: Day 20 to day 35
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Period 1: Placebo: Participants received placebo tablets twice a day (BID) in dosing period 1 (days 1 to 8).
- Period 1 Group A: OM 25 mg BID; Period 1 Group B: OM 25 mg BID: Participants received omecamtiv mecarbil 25 mg BID in dosing period 1 (days 1 to 8).
- Period 2: Placebo: Participants received placebo tablets BID in dosing period 2 (days 20 to 27).
- Period 2 Group A: OM 25 mg BID; Period 2 Group B: OM 25 mg BID: Participants received omecamtiv mecarbil 25 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Period 2 Group A: OM 37.5 mg BID: Participants received omecamtiv mecarbil 37.5 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
- Period 2 Group B: OM 50 mg BID: Participants received omecamtiv mecarbil 50 mg BID in dosing period 2 (days 20 to 27) based on their day 8 omecamtiv mecarbil Cpredose.
Arm/Group | Period 1: Placebo | Period 1 Group A: OM 25 mg BID | Period 1 Group B: OM 25 mg BID | Period 2: Placebo | Period 2 Group A: OM 25 mg BID | Period 2 Group A: OM 37.5 mg BID | Period 2 Group B: OM 25 mg BID | Period 2 Group B: OM 50 mg BID
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20 | 0/20 | 0/10 | 0/7 | 0/13 | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 2/10 | 5/20 | 3/20 | 4/10 | 3/7 | 3/13 | 1/7 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Placebo (N=10) | Period 1 Group A: OM 25 mg BID (N=20) | Period 1 Group B: OM 25 mg BID (N=20) | Period 2: Placebo (N=10) | Period 2 Group A: OM 25 mg BID (N=7) | Period 2 Group A: OM 37.5 mg BID (N=13) | Period 2 Group B: OM 25 mg BID (N=7) | Period 2 Group B: OM 50 mg BID (N=13)
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Injection site nerve damage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 2 | 1 | 3 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.